CLINICAL TRIAL: NCT07018830
Title: Multicomponent Program for Addressing Cognition in Rural Communities
Acronym: MPAAC-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-63-pbrc
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Decline
Keywords: dementia risk; rural; african american; lifestyle behavior
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent Intervention (Experimental): The multicomponent program will provide a package of altering several lifestyle behaviors simultaneously. The components will include physical activity, dietary intake, cognitive training, sleep, social engagement, and chronic disease management. The goals are to increase physical activity to the current guidelines, adhere to the Mediterranean diet, engage in cognitive training of memory, increase sleep to recommended levels, engage in social activities, and effectively manage chronic diseases.
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — Participants will be provided 11, 60 - 90 minute group sessions. They will receive behavioral strategies to address each of the lifestyle behaviors. These strategies are based on the Social Cognitive Theory and Self Determination Theory. Topics will include, but are not limited to, self-monitoring, goal setting, social support, cues, problem solving, and relapse prevention. Groups may occur both in-person and virtually.

SUMMARY:
The study is designed to develop and evaluate a multicomponent intervention program among older rural-residing and African American residents with a long-term goal of reducing risk factors for Alzheimer's disease. The motivation for this study is that previous non-pharmacological (e.g. exercise diet, social engagement) interventions have improved cognitive function in older adults with and without cognitive impairments, but these studies were largely conducted without substantial representation from residents living in rural communities or African Americans. Due to geographic, sociocultural, and environmental differences between rural residents, African Americans and other populations, it is unclear whether positive findings from previous interventions will translate to rural residents or African American individuals.

DETAILED DESCRIPTION:
It is estimated that just over 5 million Americans are currently living with Alzheimer's Disease (AD) , and that number will rise to approximately 9 million by 2050. Rural areas were shown to have 1.4 - 1.7 times higher risk of developing dementia compared to urban areas and risk was shown to be increasing in comparison to urban areas. Risk factors in rural populations include age, lower levels of education, less access to health care, and higher rates of chronic disease. The prevalence of AD among African Americans is also elevated as it is approximately double that of non-Hispanic white Americans and older African Americans may be as much as 64% more likely to develop AD compared to non-Hispanic white Americans. Some contributors to AD are similar across rural residence and African Americans, including limited health care access, lower levels of trust in physicians, limited transportation, and built environmental issues. However, to date, there are few studies that have engaged in intervention work to address reduction of AD risk factors in older adults residing in rural communities. This is particularly true for older African Americans who may face increased barriers. Therefore, there is a need to conduct more AD prevention interventions in rural communities and especially those with large proportions of African Americans.

A large literature suggests that modifiable lifestyle behaviors are associated with the risk of developing AD. For example, both cross-sectional and longitudinal studies show that lower levels of physical activity and poorer dietary intake are associated with higher risk of developing AD. African Americans have low levels of physical activity and poor dietary quality compared to corresponding non-Hispanic white Americans. Studies in cohorts with predominantly low African American representation have shown that increasing physical activity, improving dietary intake, and engaging in cognitive training, individually, have all increased cognitive test scores across multiple domains. In addition, recent data (again from predominantly white cohorts) suggests that simultaneously changing multiple of these lifestyle behaviors at the same time may engage multiple, possibly synergistic neuroprotective mechanisms and thereby maximize neuroprotective benefits.

Multicomponent interventions, or non-pharmacological interventions that address several behaviors simultaneously (e.g. physical activity, diet, cognitive training, sleep) have been shown to be effective in improving cognitive function in older adults. Recently, the two-year Finnish Geriatric Intervention study to Prevent Cognitive Impairment and Disability (FINGER) trial intervened on physical activity, diet, cognitive training, and cardiometabolic health management simultaneously; those in the intervention had significant improvements in global cognitive function, executive functioning, and processing speed, compared to a group receiving usual health care. The FINGER results were so impressive that a worldwide network of FINGER replication studies have been engaged, including the POINTER study in the United States. However, to our knowledge, none of these multicomponent studies have included a large number of rural residents or African Americans.

We will develop a multicomponent intervention specifically tailored to older adults living in rural communities, and recruit at least 20, with a maximum of 40, adults into it. The 12 session intervention will consist of group-based lifestyle change sessions at a facility determined by the community. Cognitive functioning will be assessed to determine the brain effects of the intervention in this understudied population.

Specific Aim 1: To determine if a multicomponent intervention is feasible to deliver in older rural-residing adults. Hypothesis 1: We hypothesize that the intervention will be feasible to deliver. Feasibility will be assessed through recruitment, retention, attendance, and satisfaction ratings.

Specific Aim 2: To determine if a multicomponent intervention in older rural residing adults improves cognition in the following domains: attention, processing speed, memory, and executive function. Hypothesis 2: We hypothesize that changes in all cognitive domains will improve in the interventions compared to baseline. Change over the course of the intervention will be assessed in key AD related cognitive domains (attention, processing speed, memory, and executive function).

Collecting this data sets the stage for the definitive study of the benefits of a multicomponent intervention in rural, diverse (e.g. 50% African American) residents. This will involve collecting measures of amyloid, tau, inflammation, brain metabolism, comparing findings to a control group, and assessing other AD-relevant pathways in older rural, diverse (e.g. 50% African American) adults, which could in turn increase understanding of neurobiological mechanisms and optimal physical activity recommendations for older adults residing in rural communities.

ELIGIBILITY:
Inclusion Criteria:

1. > 60 years of age
2. reside in a rural city
3. not cognitively impaired
4. physically capable of exercise
5. willing to attend group sessions
6. plan to live in the study area for the next 6 months
7. willing to allow researchers to use data for research purposes after study participation is completed
8. free of conditions that would make regular exercise unsafe as deemed by the medical investigator
9. report at least two of the following: a) no regular physical activity, b) not consuming the Mediterranean diet, 3) sleep < 6 hours per night, 4) current diagnosis of hypertension, diabetes, or obesity (by physician diagnosis or medication), 5) high school education or less, 6) history of depression.

Exclusion criteria:

1. unable or unwilling to give informed consent
2. are cognitively impaired (MMSE score of ≤ 18)
3. have sleep apnea
4. have uncontrolled hypertension (systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg).
5. have had a hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
6. have had a myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolus in the past 6 months
7. are undergoing cardiopulmonary rehabilitation
8. are currently enrolled in another randomized trial involving lifestyle or pharmaceutical interventions
9. have another member of the household that is a participant in the study
10. have plans to relocate out of the study area within the next 6 months
11. have uncontrolled diabetes that in the judgment of the MI may interfere with study participation
12. have other medical, psychiatric, or behavioral factors that in the judgment of the Principal or Medical Investigator may interfere with study participation or the ability to follow the intervention protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Study feasibility | 3 months
  Feasibility measures the likelihood of success of the study. It will be measured by a composite of 1) recruitment, 2) attendance, 3) retention, and 4) satisfaction.

SECONDARY OUTCOMES:
Mini-mental state exam | 3 months
  The Mini-mental state exam is a dementia screening tool.
Everyday Cognition Scale | 3 months
  A self- and study partner-rated questionnaire will be used to measure cognitive change over time in overall functional ability.
Wide Range Achievement Test - Reading Subtest | 3 months
  Reading level will be assessed using a test of irregular word reading that assesses participant's ability to recognize and pronounce words in isolation
Auditory Verbal Learning Test | 3 months
  A delayed recall test will be used to assess cognitive function.
Cultural Consensus Modeling | 3 months
  A multi-method approach to identify shared cultural beliefs around a specific subject.
Mediterranean diet screener | 3 months
  This 14-item questionnaire assesses adherence to the Mediterranean diet.
Perceived Sleep Quality Index | 3 months
  The PSQI is a measure of subjective sleep duration and quality over a 4-week period. It is the most widely used validated sleep questionnaire in the field.
Physical Activity Readiness Questionnaire | 3 months
  The PAR-Q+ is a seven-question pre-participation screening tools for physical activity.
Short Physical Performance Battery | 3 months
  The SPPB is a brief performance battery based on timed short distance walk, repeated chair stands and balance test.
Community Healthy Activities Model Program for Seniors | 3 months
  The questionnaire assesses the weekly frequency and duration of various physical activities typically undertaken by older adults.
Height | 3 months
  Height will be measured using a standard stadiometer.
Weight | 3 months
  Weight will be measured using a standard stadiometer and scale.
Blood Pressure | 3 months
  Blood pressure will be measured by trained staff using electronic and/or manual blood pressure machine.
Health Related Quality of Life | 3 months
  The HRQL measures health related quality of life.
Geriatric Depression Scale | 3 months
  The GDS is a measure of depression that is able to discriminate the pattern of depressive symptoms from the general characteristics of the elderly population.
The Food Noise Questionnaire | 3 months
  The Food Noise Questionnaire (FNQ) provides a brief 5-item practical tool for researchers and clinicians to measure food noise.
Lubben Social Network Scale | 3 months
  The questionnaire screens for social isolation through assessment of social networks and social supports.
Treatment satisfaction | 3 months
  Participants will complete a satisfaction questionnaire adapted from the investigators' previous study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Newton, Jr, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data can be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available June 2026
Access Criteria: All study data will be available. Request from the investigative team.